CLINICAL TRIAL: NCT00362089
Title: The Impact of the Nutritional Fatty Acids During Pregnancy and Lactation for Early Human Adipose Tissue Development
Brief Title: Fatty Acids During Pregnancy and Lactation and Body Fat Mass in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Else Kröner-Fresenius-Foundation; International Unilever-Foundation; Danone Research (Unknown); EU funding by EARNEST consortium;German Ministry of Education and Research GF-GFGI01120708) (Unknown)
Responsible Party: Principal Investigator, Ulrike Amann-Gassner, PhD, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EKFZ001_CN; INFAT (Other: Else Kroener-Fresenius-Center for Nutritional Medicine)
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Overweight; Obesity
Keywords: n-3 fatty acids; n-6 fatty acids; long chain polyunsaturated fatty acids; pregnancy; lactation; breast feeding; breast milk; adipose tissue; newborn; fetal development
MeSH Terms: conditions — Overweight; Obesity; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Marinol (Active Comparator): Intervention group with Marinol D40 fish oil capsules
  Interventions: Dietary Supplement: Marinol D-40
- Nutrition counseling (No Intervention): Control group

INTERVENTIONS:
Dietary Supplement: Marinol D-40 — Marinol D-40, three capsules per day, from 15th week of gestation until 4th month of lactation
  Arms: Marinol

SUMMARY:
Pregnant and lactating women receive n-3 fatty acids starting from week 15 of gestation until 4 months post-partum (pp) in comparison to a control group, who only gets information about adequately healthy nutrition during pregnancy and lactation.

The amount of fat in newborns is measured through skinfold thickness, ultrasound, and magnetic resonance imaging (MRI).

It is hypothesised that a reduction in arachidonic acid intake and an increase of n-3 LC PUFAs (long chain polyunsaturated fatty acids) via supplements containing docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA) could lead to less expansive fat tissue development in the first year of life.

DETAILED DESCRIPTION:
The prevalence of overweight and obese children and adolescents dramatically increased during the last two decades. In Germany every 5th school child is overweight and 4 - 8% of all children are obese.

Recent studies suggest that fatty acids in maternal nutrition may have an impact on the fat tissue development during the fetal period.

Animal studies showed that a reduction in the arachidonic acid intake, a higher intake of n-3 LC PUFAs (i.e. DHA and EPA) and a resulting lower n-6/n-3 fatty acid ratio in food will cause less expansive fat tissue development in the first year of life.

In vitro studies and personal observations in animal studies also showed that n-6 fatty acids (i.e. arachidonic acid) stimulate the differentiation of preadipocytes to adipocytes whereas n-3 fatty acids (i.e. DHA and EPA) have the contrary effect.

The impact of the maternal fatty acid pattern on the early fat tissue development can only be clarified in an intervention study.

Therefore it is planned to recruit 204 pregnant women in the 14th week of gestation. They will be randomly assigned to the intervention or control group.

The intervention group will receive n-3 LC-PUFAs (DHA and EPA) as fish oil capsules from the 15th week of gestation until 4 months pp, the control group will get nutrition counselling according to the recommendations of the German Society for Nutrition during the same time period. Blood samples of the pregnant and lactating women, umbilical cord blood, placental tissue and blood of the newborns will be collected for fatty acid analysis.

Body fat mass in newborns will be determined from delivery until 4 months pp via skinfold measurement, ultrasound, and MRI.

The hypothesis is that newborns in the group of the "supplemented" mothers will have less expansive fat tissue development than children from mothers in the control group.

This would be an innovative primary preventive approach in a period of increasing prevalence of overweight and obese children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <= 15th week of gestation
* Age: 18-43 years
* Written informed consent
* Body mass index (BMI) before pregnancy between 18 and 30 km/m2

Exclusion Criteria:

* High risk pregnancy
* Hypertonus
* Chronic diseases (i.e. diabetes mellitus)
* Psychiatric diseases
* Former supplementation with LC-PUFA

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2006-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
amount of fat mass in the offspring | at birth, 6 weeks, 4 months, 1 year postpartum
  skinfold thickness measurements

SECONDARY OUTCOMES:
amount of fat mass in the offspring | at 1,5 years, 2 years, 2.5 years, 3 years, 4 years and 5 years postpartum (follow-up)
  skinfold thickness measurements
offspring body height | at birth, 6 weeks, 4 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years, 4 years and 5 years postpartum
head circumference of newborns, infants and children | at birth, 6 weeks, 4 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years, 4 years and 5 years postpartum
blood lipids of pregnant and lactating women | 15th wk gestation, 32nd wk gestation, 6 weeks pp, 4 months pp
fatty acid profile of phospholipids and erythrocyte membrane lipids, fatty acid metabolites | 15th wk gestation, 32nd wk gestation, birth, 6 wks, 4 months, 1 year, 3 years postpartum
  maternal and offspring blood cells and plasma, placenta, umbilical cord tissue, blood cells and plasma, breast milk
daily intake of maternal fatty acids | 15 wks gestation, 32nd wks gestation, 6 wks pp
  7 day dietary records
offspring abdominal subcutaneous and preperitoneal fat | 6 weeks, 4 months , 1 year , 1.5 years , 2 years, 2.5 years, 3 years, 4 years, 5 years postpartum
  Ultrasonography
offspring fat mass, abdominal fat | 6 weeks, 4 months, 5 years postpartum
  magnetic resonance imaging
maternal and offspring gene expression (mRNA, miRNA) | 15 wk gestation, 32nd wk gestation (maternal), birth, 3 years (offspring)
  placenta, umbilical cord tissue, white blood cells, blood plasma
maternal and offspring DNA analysis (SNPs, DNA methylation) | 15 wk gestation, 32nd wk gestation (maternal), birth, 3 years (offspring)
  placenta, umbilical cord tissue, white blood cells
epigenetic analyses (histone modification, DNA methylation) | birth
  placenta, umbilical cord tissue, white blood cells
cytokines, adipokines and hormone analysis | 15th wk gestation, 32nd wk gestation, 6 wks pp, 4 months pp (maternal), birth, 4 months, 1 year, 3 years postpartum (offspring)
  maternal and offspring blood cells and plasma, placenta, umbilical cord blood cells and plasma, breast milk
protein analysis, proteomics | 15th wk gestation, 32nd wk gestation (maternal), birth, 4 months, 1 year, 3 years postpartum (offspring)
  maternal and offspring blood cells and plasma, placenta, umbilical cord blood cells and plasma
metabolomics, lipidomics | 15th wk gestation, 32nd wk gestation (maternal), birth, 4 months, 1 year, 3 years postpartum (offspring)
  maternal and offspring blood cells and plasma, placenta, umbilical cord blood cells and plasma
breast milk oligosaccharides | 6 wks and 4 months postpartum
offspring atopic eczema | 1.5 years - 5 years postpartum
  parent questionnaire
offspring allergic diseases (asthma, rhinitis) | 5 years postpartum
  parent questionnaire
developmental evaluation of children | 2 years - 5 years postpartum
  parent questionnaire (based on Minnesota Scales)
motor development of children | 4 years and 5 years postpartum
physical activity of children | 2 years - 5 years postpartum
  parent questionnaire
dietary intake of children | 2 years - 5 years postpartum
  3 day dietary record
offspring body weight | at birth, 6 weeks, 4 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years, 4 years and 5 years postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Hans Hauner, Prof., Principal Investigator — Else Kröner-Fresenius-Zentrum für Ernährungsmedizin, Technische Universität München
Locations (1):
- Else Kröner-Fresenius-Zentrum für Ernährungsmedizin, Technische Universität München, Munich, Germany

REFERENCES:
- [Background] Hauner H, Vollhardt C, Schneider KT, Zimmermann A, Schuster T, Amann-Gassner U. The impact of nutritional fatty acids during pregnancy and lactation on early human adipose tissue development. Rationale and design of the INFAT study. Ann Nutr Metab. 2009;54(2):97-103. doi: 10.1159/000209267. Epub 2009 Mar 19. PMID 19295192
- [Background] Much D, Brunner S, Vollhardt C, Schmid D, Sedlmeier EM, Bruderl M, Heimberg E, Bartke N, Boehm G, Bader BL, Amann-Gassner U, Hauner H. Effect of dietary intervention to reduce the n-6/n-3 fatty acid ratio on maternal and fetal fatty acid profile and its relation to offspring growth and body composition at 1 year of age. Eur J Clin Nutr. 2013 Mar;67(3):282-8. doi: 10.1038/ejcn.2013.2. Epub 2013 Jan 23. PMID 23340492
- [Background] Brunner S, Schmid D, Huttinger K, Much D, Bruderl M, Sedlmeier EM, Kratzsch J, Amann-Gassnerl U, Bader BL, Hauner H. Effect of reducing the n-6/n-3 fatty acid ratio on the maternal and fetal leptin axis in relation to infant body composition. Obesity (Silver Spring). 2014 Jan;22(1):217-24. doi: 10.1002/oby.20481. Epub 2013 Sep 10. PMID 23596009
- [Background] Much D, Brunner S, Vollhardt C, Schmid D, Sedlmeier EM, Bruderl M, Heimberg E, Bartke N, Boehm G, Bader BL, Amann-Gassner U, Hauner H. Breast milk fatty acid profile in relation to infant growth and body composition: results from the INFAT study. Pediatr Res. 2013 Aug;74(2):230-7. doi: 10.1038/pr.2013.82. Epub 2013 May 28. PMID 23715519
- [Background] Brunner S, Schmid D, Huttinger K, Much D, Heimberg E, Sedlmeier EM, Bruderl M, Kratzsch J, Bader BL, Amann-Gassner U, Hauner H. Maternal insulin resistance, triglycerides and cord blood insulin in relation to post-natal weight trajectories and body composition in the offspring up to 2 years. Diabet Med. 2013 Dec;30(12):1500-7. doi: 10.1111/dme.12298. Epub 2013 Sep 11. PMID 23909286
- [Result] Hauner H, Much D, Vollhardt C, Brunner S, Schmid D, Sedlmeier EM, Heimberg E, Schuster T, Zimmermann A, Schneider KT, Bader BL, Amann-Gassner U. Effect of reducing the n-6:n-3 long-chain PUFA ratio during pregnancy and lactation on infant adipose tissue growth within the first year of life: an open-label randomized controlled trial. Am J Clin Nutr. 2012 Feb;95(2):383-94. doi: 10.3945/ajcn.111.022590. Epub 2011 Dec 28. PMID 22205307
- [Derived] Meyer DM, Brei C, Stecher L, Brunner S, Hauner H. Maternal insulin resistance, triglycerides and cord blood insulin are not determinants of offspring growth and adiposity up to 5 years: a follow-up study. Diabet Med. 2018 Oct;35(10):1399-1403. doi: 10.1111/dme.13765. Epub 2018 Aug 2. PMID 29938825
- [Derived] Meyer DM, Brei C, Stecher L, Much D, Brunner S, Hauner H. The relationship between breast milk leptin and adiponectin with child body composition from 3 to 5 years: a follow-up study. Pediatr Obes. 2017 Aug;12 Suppl 1:125-129. doi: 10.1111/ijpo.12192. Epub 2016 Nov 10. PMID 27863153
- [Derived] Brei C, Stecher L, Much D, Karla MT, Amann-Gassner U, Shen J, Ganter C, Karampinos DC, Brunner S, Hauner H. Reduction of the n-6:n-3 long-chain PUFA ratio during pregnancy and lactation on offspring body composition: follow-up results from a randomized controlled trial up to 5 y of age. Am J Clin Nutr. 2016 Jun;103(6):1472-81. doi: 10.3945/ajcn.115.128520. Epub 2016 Apr 6. PMID 27053380
- [Derived] Brei C, Much D, Heimberg E, Schulte V, Brunner S, Stecher L, Vollhardt C, Bauer JS, Amann-Gassner U, Hauner H. Sonographic assessment of abdominal fat distribution during the first year of infancy. Pediatr Res. 2015 Sep;78(3):342-50. doi: 10.1038/pr.2015.108. Epub 2015 Jun 8. PMID 26053137
- [Derived] Brunner S, Schmid D, Zang K, Much D, Knoeferl B, Kratzsch J, Amann-Gassner U, Bader BL, Hauner H. Breast milk leptin and adiponectin in relation to infant body composition up to 2 years. Pediatr Obes. 2015 Feb;10(1):67-73. doi: 10.1111/j.2047-6310.2014.222.x. Epub 2014 Apr 14. PMID 24729519